CLINICAL TRIAL: NCT01886079
Title: The Effects of Dexmedetomidine on Postoperative Renal Function in Valvular Heart Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4-2013-0194
Record Dates: First submitted 2013-06-18; First posted 2013-06-25 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Dexmedetomidine group (Experimental)
  Interventions: Drug: dexmedetomidine
- Saline group (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: dexmedetomidine — 0.4 mcg/kg/h, IV, The infusion of study drug is started after anesthesia induction and continued until 24 hours after surgery
  Arms: Dexmedetomidine group
Drug: Saline — 0.4 mcg/kg/h, IV
  Arms: Saline group

SUMMARY:
The purpose of study is to compare the incidence of acute kidney injury in patients receiving perioperative dexmedetomidine or placebo undergoing valvular heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* adult patients over the age of 20 scheduled for valvular heart surgery

Exclusion Criteria:

* Left ventricular-ejection fraction < 30%
* Preexisting congestive heart failure
* Severe coronary artery disease
* Hemodynamically unstable arrhythmia
* Cardiogenic shock during perioperative period
* Ventricular assist device
* Severe renal dysfunction (eGFR < 15ml/min per 1.73m2)

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Comparison of postoperative renal function in patients with or without dexmedetomidine undergoing valvular heart surgery: | 24 hours after surgery.
  BUN/Creatinine, cystatin C, eGFR, urine output Incidence of acute kidney injury (based on the AKIN criteria)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea